CLINICAL TRIAL: NCT00579293
Title: Development of a Computer Assisted Survivor Screening For Adult Survivors of Childhood Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Jennifer Ford, PhD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 04-098
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2008-07-28 (Estimated); Status verified 2008-07

CONDITIONS: Childhood Cancer
Keywords: adult survivor of childhood cancer; computer assisted screening of survivors (CASS)
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
This study will compare two ways of having people respond to a questionnaire about health and emotional well-being: on a computer and with paper and pencil. We will see how long it takes using both methods. We will also ask you how you feel about using a computer to answer the questions.

DETAILED DESCRIPTION:
To determine feasibility of using the Computer Assisted Survivor Screening (CASS) as a routine screening measure for the survivor population. Specifically, to determine patient acceptance, time to completion, and burden associated with the CASS. To examine the potential utility of the CASS as a routine screening measure in the survivor population. To validate the CASS against the SCL-90-R screening measure. Calculate the sensitivity,specificity, positive and negative predictive values, diagnostic agreement and ROC curve of the CASS compared to the SCL-90. Determine the optimal cut-off scores to optimize agreement between the CASS and the SCL-90.

ELIGIBILITY:
Inclusion Criteria:

* Currently at least 18 years of age and not older than 49 years of age
* Diagnosed with first malignancy before the age of 22
* Completed all cancer treatment at least three years prior
* Able to complete the survey instruments in English
* Scheduled for a routine off-treatment follow-up oncology appointment
* Currently disease-free and not receiving any cancer treatment

Exclusion Criteria:

* History of a central nervous system tumor
* A sensory or cognitive impairment that would interfere with completion of the survey
* Currently undergoing treatment by a psychiatrist or psychologist (ie., currently receiving psychotherapy and/or psychotropic medications, as per self-report)

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: adult survivors of childhood cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2004-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ford, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org